CLINICAL TRIAL: NCT04842513
Title: Multi Peptide Vaccination with Pam3Cys-GDPKHPKSF (XS15) As an Immunomodulator in Addition to Standard Postoperative Radiation Therapy and Temozolomide Chemotherapy in Newly Diagnosed HLA-A2-positive MGMT-methylated Glioblastoma
Brief Title: Multi Peptide Vaccination with XS15 in Addition to Standard Postoperative Radiation Therapy and Temozolomide Chemotherapy in Newly Diagnosed Glioblastoma
Acronym: GLIO-XS15
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003357-30
Record Dates: First submitted 2021-03-01; First posted 2021-04-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2023-12

CONDITIONS: Glioblastoma Multiforme of Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multipeptide plus XS15 (Experimental): The vaccine will be applied by subcutaneous injection into the abdominal skin of the study patient. Vaccination will take place monthly (V1, V2 and V3). A total of three vaccinations will be performed. Peptide vaccines should be injected into the skin at the lower part of the abdomen of the patients. The exact site of vaccination (right or left) will be determined at the time of first vaccination and should not be changed during subsequent vaccinations.
  Interventions: Drug: Multipeptide plus XS15

INTERVENTIONS:
Drug: Multipeptide plus XS15 — The vaccine will be applied by subcutaneous injection into the abdominal skin of the study patient. Vaccination will take place monthly (V1, V2 and V3). A total of three vaccinations will be performed. Peptide vaccines should be injected into the skin at the lower part of the abdomen of the patients. The exact site of vaccination (right or left) will be determined at the time of first vaccination and should not be changed during subsequent vaccinations.

SUMMARY:
Newly diagnosed HLA-A2-positive MGMT-methylated glioblastoma patients will be vaccinated with a Multi peptide vaccination with Pam3Cys-GDPKHPKSF (XS15) as an immunomodulator in addition to standard postoperative radiation therapy and temozolomide chemotherapy to assess immunogenicity, efficacy, safety of the combination of multipeptide vaccination and the immune modulator XS15 emulsified in Montanide ISA 51 VG

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be considered for admission to the trial:

For screening phase: (Consent C1)

1. .Must be ≥ 18 years at the time of signing the informed consent 2. Suspected Glioblastoma (presenting with a MRI suggestive of glioblastoma and eligible for gross or subtotal resection and standard radiotherapy with temozolomide) For Vaccination phase (Consent C2)

1. Histologically confirmed, newly diagnosed IDH1-wildtype glioblastoma (astrocytoma WHO grade IV)
2. MGMT gene promoter methylation
3. HLA phenotype HLA-A*02:01 (as determined by a PCR-based 4-digit typing method)
4. Gross or subtotal resection (20%, as determined by MRI)
5. Postoperative MRI
6. KPS ≥70%
7. Life expectancy > 6 months
8. Patient is a candidate for and willing to receive standard radiation therapy with TMZ followed by maintenance TMZ cycles
9. Patient is not on steroids or on stable or decreasing steroid levels not exceeding 2 mg/day dexamethasone (or equivalent doses of other steroids) during the last 3 days prior to first dose of IMP (Vaccination 1)
10. Absolute lymphocyte count (ALC) >0.5 x109/L (re-screening of lymphocyte counts is allowed at day of vaccination)
11. Ability of subject to understand and the willingness to sign written informed consent for study participation prior to any study related assessments/procedures. Able to adhere to the study visit schedule and other protocol requirements.
12. Female Patient of childbearing potential1 and male patients with female partner of childbearing potential1 is willing to use highly effective contraceptive methods during treatment and for 30 days after the end of treatment. According to the CTFG Recommendations highly effective contraceptive methods are:

    * combined hormonal contraceptive associated with inhibition of ovulation (oral,-intravaginal,-transdermal)
    * progestogen-only hormonal contraception associated with inhibition of ovulation (pral injectable, implantable)
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system (IUS)
    * bilateral tubal occlusion,
    * vasectomized partner2,
    * sexual abstinence3.
13. Negative Covid 19 Quick Test
14. Female subjects must abstain from breastfeeding during study participation and 30 days after study drug discontinuation.
15. Male subjects must refrain from donating semen or sperm while on study
16. All subjects must agree to refrain from donating blood while on study drug and for 30 days after discontinuation from this study treatment.
17. All subjects must agree not to share medication.

Exclusion Criteria:

* Subjects presenting with any of the following criteria will not be included in the trial:

  1. Karnofsky performance score (KPS) < 70%
  2. Patient who cannot undergo MRI assessments
  3. Only Biopsy available
  4. Women during pregnancy and lactation.
  5. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
  6. Participation in other clinical trials or observation period of competing trials.
  7. Platelet count decrease < 75 x109/L
  8. Bilirubin > 1.5 x ULN (upper limit of normal according to the performing lab's reference range)
  9. ALT4 > 3 x ULN
  10. AST5 > 3 x ULN
  11. GGT > 2.5 x ULN
  12. Serum creatinine increased > 1.5 x ULN
  13. HIV infection or active Hepatitis B or C infection, or active infections requiring oral or intravenous antibiotics or that can cause a severe disease and pose a severe danger to lab personnel working on patients' blood or tissue (e.g. rabies).
  14. Prior therapy for glioma (except surgery and steroids) including but not limited to carmustine wafers and immunotherapy. Note: History of low grade glioma that did not require prior treatment with chemotherapy or radiotherapy is not an exclusion criterion.
  15. Clinically relevant autoimmune diseases (with the exception of thyroid diseases).
  16. Immunosuppression, not related to prior treatment for malignancy, or prior drug reaction
  17. Other vaccinations with active or attenuated viruses should be restricted during the peptide vaccination period.
  18. Enzyme-inducing antiepileptic drugs
  19. Patients with prior stem cell transplantation or solid organ transplantation.
  20. Any condition that in the judgment of the investigator interferes with the probability that an individual patient may receive and benefit from APVAC vaccinations (e.g. high risk of early disease progression / recurrence; immunocompromised status; anticipated compliance problems)
  21. Serious illness or condition, which according to the investigator, poses an undue risk for the patient when participating in the trial, including, but not limited to, any of the following:

      * Clinically symptomatic cardiovascular disease:(New York Heart Association class III-IV congestive heart failure)
      * Symptomatic peripheral vascular disease (Definition z.B. > Stage III)
      * Severe pulmonary dysfunction (Definition: z.B. requirement for oxygen supplement
      * Severe diabetes
      * History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 5 years unless the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Adevrse Events | at 12 months after last vaccination
  The assessment of safety of the IMP will be accomplished by documentation of adverse events and grading according to CTCAE from first vaccination throughout the end of treatment, until 30 days after last vaccination.
Change of immunogenicity parameter from baselien | at 30 days, 60 days and 90 days from first vaccination and at 12 months after last vaccination
  The assessment of immunogenicity is the central biological efficacy endpoint of the clinical trial. Measurements of the induction of T-cell response after vaccination at 30 days, 60 days and 90 days from first vaccination and at 12 months after last vaccinationcompared to baseline as determined by ELISpot

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Tabatabai, Prof, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No